CLINICAL TRIAL: NCT02566928
Title: Patient-Centered Comparative Effectiveness Research (CER) Study of Home-based Interventions to Prevent CA-MRSA Infection Recurrence
Acronym: CAMP-2
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Clinical Directors Network (Network)
Collaborators: Rockefeller University (Other); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CER-1402-10800
Record Dates: First submitted 2015-09-30; First posted 2015-10-02 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Methicillin-Resistant Staphylococcus Aureus; Recurrence; Staphylococcal Skin Infections; Antibiotic Resistance
Keywords: Methicillin-Resistant Staphylococcus aureus; Recurrence; Practice Based Research Network; Community Health Workers/Promotoras; Decolonization and Decontamination; Staphylococcal Skin Infections; Household Transmission
MeSH Terms: conditions — Recurrence; Staphylococcal Skin Infections | interventions — Bacitracin; Mupirocin; chlorhexidine gluconate

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Decolonization and Decontamination (Experimental): Index Patients will receive: 1) guidelines-directed care, which may consist of incision, drainage, oral antibiotics, and antibiogram-based antibiotic prescribing, and 2) a home-based intervention implemented by Community Health Workers/Promotoras that includes index patient and household member education and instructions to complete a decolonization and decontamination regimen, along with printed materials describing a standard hygiene protocol for reducing household contamination. Index patients and consenting household members will complete a decolonization regimen consisting of twice-daily application of 2% mupirocin ointment to the anterior nares with a clean cotton applicator for five days, as well as daily bathing with chlorhexidine wash for five days. The household decontamination hygiene protocol includes the use of hand-washing, surface disinfection, and laundering.
  Interventions: Drug: 2% mupirocin ointment; Other: Chlorhexidine wash; Behavioral: Hygiene protocol
- Usual Care (No Intervention): Index Patients will receive: 1) guidelines-directed care, which may consist of incision, drainage, and oral antibiotics, as well as antibiogram-based antibiotic prescribing, and 2) printed materials describing a standard hygiene protocol for reducing household contamination.

INTERVENTIONS:
Drug: 2% mupirocin ointment — Index patients and consenting household members will complete a decolonization regimen consisting of twice-daily application of mupirocin ointment to the anterior nares with a sterile cotton applicator for five days.
  Other Names: Bacitracin; Bactroban
  Arms: Decolonization and Decontamination
Other: Chlorhexidine wash — Index patients and consenting household members will daily daily for five days with chlorhexidine wash.
  Other Names: Hibiclens
  Arms: Decolonization and Decontamination
Behavioral: Hygiene protocol — Index patients and consenting household members will be given educational materials and instructed to in the use of hand-washing, surface disinfection, and laundering.
  Arms: Decolonization and Decontamination

SUMMARY:
The overall goal of the project is to develop and evaluate a home-based intervention to prevent re-infection and transmission of Community-Acquired Methicillin-resistant Staphylococcus aureus (CA-MRSA) in patients presenting to primary care with skin or soft tissue infections (SSTIs). Centers for Disease Control (CDC) CA-MRSA guidelines include incision and drainage, antibiotic sensitivity testing and antibiogram-directed prescribing. Re-infections are common, ranging from 16% to 43%, and present significant challenges to clinicians, patients and their families. Several decolonization and decontamination interventions have been shown to reduce Hospital-Acquired MRSA (HA-MRSA) re-infection and transmission in intensive care units. Few studies examine the feasibility and effectiveness of these infection prevention interventions into primary care settings, and none employ Community Health Workers (CHWs) or "promotoras" to provide home visits for education and interventions about decolonization and decontamination. This comparative effectiveness research/patient centered outcomes research builds upon a highly stakeholder-engaged community-academic research and learning collaborative, including practicing clinicians, patients, clinical and laboratory researchers, and barbers/beauticians. Clinical Directors Network (CDN), an established, NIH-recognized best practice Federally Qualified Health Center (FQHC) Practice-based Research Network (PBRN), and The Rockefeller University propose to address this question through the completion of four aims: (1) To evaluate the comparative effectiveness of a CHW/Promotora-delivered home intervention (Experimental Group) as compared to Usual Care (Control Group) on the primary patient-centered and clinical outcome (SSTI recurrence rates) and secondary patient-centered and clinical outcomes (pain, depression, quality of life, care satisfaction) using a two-arm randomized controlled trial (RCT). (2) To understand the patient-level factors (CA-MRSA infection prevention knowledge, self-efficacy, decision-making autonomy, prevention behaviors/adherence) and environmental-level factors (household surface contamination, household member colonization, transmission to household members) that are associated with differences in SSTI recurrence rates. (3) To understand interactions of the intervention with bacterial genotypic and phenotypic variables on decontamination, decolonization, SSTI recurrence, and household transmission. (4) To explore the evolution of stakeholder engagement and interactions among patients and other community stakeholders with practicing community-based clinicians and academic laboratory and clinical investigators over the duration of the study period.

ELIGIBILITY:
Inclusion Criteria:

* between 7 to 70 years of age
* fluent in English or Spanish
* plans to receive care in the Community Health Center during the next year
* presents with signs and symptoms of a SSTI
* willing/able to provide informed consent

Exclusion Criteria:

* The patient is unwilling to provide informed consent
* acutely sick (for example, crying, wheezing, bleeding, screaming or shaken)
* unable to participate in a discussion about the study

Ages: 7 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 278 (Estimated)
Dates: Start 2015-10; Primary Completion 2018-11 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
SSTI Recurrence Rate | 3 months
  Defined as having one or more discrete clinical SSTIs at the same or new site in addition to the baseline infection. Defined by self-report and review of patients' medical records for evidence of one or more of the following: (1) new SSTIs for which the patient presents for medical care, (2) the initial SSTI which failed to heal despite treatment (including I&D and/or antibiotic prescription), (3) a new laboratory-confirmed culture of MRSA or Methicillin Sensitive Staphylococcus aureus (MSSA).
SSTI Recurrence Rate | 6 months
  Defined as having one or more discrete clinical SSTIs at the same or new site in addition to the baseline infection. Defined by self-report and review of patients' medical records for evidence of one or more of the following: (1) new SSTIs for which the patient presents for medical care, (2) the initial SSTI which failed to heal despite treatment (including I&D and/or antibiotic prescription), (3) a new laboratory-confirmed culture of MRSA or Methicillin Sensitive Staphylococcus aureus (MSSA).
SSTI Recurrence Rate | 12 months
  Defined as having one or more discrete clinical SSTIs at the same or new site in addition to the baseline infection. Defined by self-report and review of patients' medical records for evidence of one or more of the following: (1) new SSTIs for which the patient presents for medical care, (2) the initial SSTI which failed to heal despite treatment (including I&D and/or antibiotic prescription), (3) a new laboratory-confirmed culture of MRSA or Methicillin Sensitive Staphylococcus aureus (MSSA).

SECONDARY OUTCOMES:
Clinical Response Questionnaire | 1, 3, 6, and 12 months
Subsequent SSTI Self-Report | 1, 3, 6, and 12 months
Medication Adherence Scale | 1, 3, 6, and 12 months
Satisfaction with Participating in Social Roles | Baseline, 3, 6, and 12 months
Depression Short Form | Baseline, 3, 6, and 12 months
Pain Interference Short Form | Baseline, 3, 6, and 12 months
Short Form 36 Health Survey | Baseline, 3, 6, and 12 months
Hygiene Score | Baseline, 1, 3, 6, and 12 months
Household Crowding Index | Baseline and 3 months
Number of participants with adverse events | Baseline, 1, 3, 6, and 12 months
Incidence of Mupirocin Resistance | Baseline and 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan N Tobin, PhD, Principal Investigator — Clinical Directors Network
Locations (6):
- United States (6):
  - NYU Lutheran Family Health Centers, Brooklyn, New York
  - NYU Lutheran Medical Center Emergency Department, Brooklyn, New York
  - Coney Island Hospital, Brooklyn, New York
  - Community Healthcare Network, New York, New York
  - Metropolitan Hospital Center, New York, New York
  - Urban Health Plan, The Bronx, New York

REFERENCES:
- [Derived] D'Orazio B, Ramachandran J, Khalida C, Gonzalez J, Kost RG, Vasquez KS, Evering TH, Holder T, Hassen GW, Hammock R, Nguyen R, Davis R, Millan K, Johnson V, Parola C, Coller BS, Tobin JN. Stakeholder Engagement In a Comparative Effectiveness/Implementation Study to Prevent Staphylococcus Aureus Infection Recurrence: CA-MRSA Project (CAMP2). Prog Community Health Partnersh. 2022;16(1):45-60. doi: 10.1353/cpr.2022.0005. PMID 35342110